CLINICAL TRIAL: NCT00648336
Title: Single-Dose Fasting In Vivo Bioequivalence Study of Mercaptopurine (50 mg; Mylan) and Purinethol® Tablets (50 mg; Gate) in Healthy Male Volunteers
Brief Title: Fasting Study of Mercaptopurine 50 mg and Purinethol® Tablets 50 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MERC-0360
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Mercaptopurine

ARMS (2):
- 1 (Experimental): Mercaptopurine 50 mg
  Interventions: Drug: Mercaptopurine 50 mg
- 2 (Active Comparator): Purinethol® Tablets 50 mg
  Interventions: Drug: Purinethol® Tablets 50 mg

INTERVENTIONS:
Drug: Mercaptopurine 50 mg — 50mg, single dose fasting
  Arms: 1
Drug: Purinethol® Tablets 50 mg — 50mg, single dose fasting
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's mercaptopurine 50 mg tablets to Gate's Purinethol® 50 mg tablets following a single, oral 50 mg (1 x 50 mg) dose administered under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older.
2. Sex: Male
3. Volunteers are to be sterile (documentation required) or during the course of the study, from study screen until 3 months after study exit, non-sterile male volunteers must use a spermicide-containing barrier method of contraception to prevent the pregnancy of their sexual partner. This advice should be documented in the informed consent form.
4. Weight: At least 60 kg (132 lbs.) and within 15% of Ideal Body Weight (IBW), as referenced by the Table of ""Desirable Weights of Adults"" Metropolitan Life Insurance Company, 1999 (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
5. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, laboratory evaluation, 12-lead ECG, hepatitis B and hepatitis C tests, HIV test, and urine drug screen including amphetamine, barbiturates, benzodiazepine, cannabinoid, cocaine, opiate screen, phencyclidine, and methadone) performed within 14 days of the initial dose of study medication.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco products within 1 year of the start of the study.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamin or herbal supplements within 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. History of drug and/or alcohol abuse within 1 year of the start of the study.
   6. A positive result for any drug in the urine drug screen.
3. Medications:

   1. Use of any medication within the 14 days prior to the initial dose of study medication.
   2. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
   3. Use of allopurinol or aminosalicylates (e.g. olsalazine, mesalamine, sulfasalazine) within 3 months of the start of the study.
4. Diseases:

   1. History of any significant chronic disease and/or hepatitis.
   2. Acute illness at the time of either the pre-study medical evaluation or dosing.
   3. A positive HIV, hepatitis B, or hepatitis C test.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
   3. Abnormal liver function tests (i.e. ALT (SGPT), AST (SGOT), alkaline phosphatase, bilirubin).
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to mercaptopurine or other related products.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration.
11. Family history of a deficiency in the enzyme thiopurine methyltransferase.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-11; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D., Principal Investigator — PRACS Institute Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html